CLINICAL TRIAL: NCT01905683
Title: Open-label, Non-controlled, Multicenter Long-term Study to Investigate the Safety and Efficacy of Xeomin® (Incobotulinumtoxin A, NT 201) for the Treatment of Spasticity of the Lower Limb(s) or of Combined Spasticity of Upper and Lower Limb in Children and Adolescents (Age 2 - 17 Years) With Cerebral Palsy
Brief Title: Long-term Open-label Study of Botulinumtoxin Type A to Treat Spasticity of Leg(s) or Leg(s) and Arm in Cerebral Palsy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merz Pharmaceuticals GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MRZ60201_3071_1; 2012-005055-17 (EudraCT Number)
Record Dates: First submitted 2013-07-18; First posted 2013-07-23 (Estimated); Results first posted 2017-10-27 (Actual); Last update posted 2017-10-27 (Actual); Status verified 2017-09

CONDITIONS: Lower Limb and Combined Lower Limb and Upper Limb Spasticity Due to Cerebral Palsy
MeSH Terms: interventions — incobotulinumtoxinA; Botulinum Toxins, Type A

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 16-20 Units per kg body weight incobotulinumtoxinA (Experimental)
  Interventions: Drug: IncobotulinumtoxinA (16-20 Units per kg body weight)

INTERVENTIONS:
Drug: IncobotulinumtoxinA (16-20 Units per kg body weight) — Active ingredient: Clostridium Botulinum neurotoxin type A free from complexing proteins. Solution for injection prepared by reconstitution of powder with 0.9% Sodium Chloride (NaCl); Total dose per injection cycle: up to 500 units; Mode of administration: intramuscular injection into spastic muscles.
  Other Names: Xeomin; NT 201; Botulinum toxin type A (150 kiloDalton), free from complexing proteins

SUMMARY:
The purpose of this study is to determine whether injections of Botulinum toxin type A into muscles of the leg(s) or of leg(s) and one arm are safe in treating children/adolescents (age 2-17 years) long-term with increased muscle tension/uncontrollable muscle stiffness (spasticity) due to cerebral palsy.

ELIGIBILITY:
Inclusion Criteria:

Main clinical inclusion criteria for completers of study MRZ60201_3070_1:

* Subject with lower limb [LL] spasticity who completed lead-in study MRZ60201_3070_1 in any of the three dose groups with duration of both injection cycles between 12 and 16 weeks.
* Ashworth scale [AS] score ≥2 in plantar flexors (at least unilaterally). For subjects with an AS score of 1, the investigator has to decide on the clinical need for reinjection.
* Clinical need for spasticity treatment with NT 201 according to the clinical judgment of the investigator for:

Unilateral treatment of LL spasticity with 8 U/kg BW NT 201 (maximum of 200 U) into pes equinus and need for additional 8 U/kg BW NT 201 (maximum of 200 U) for treatment of clinical pattern flexed knee or adducted thigh (ipsilateral) or bilateral treatment of LL spasticity with 8 U/kg BW NT 201 (maximum of 200 U) into pes equinus on each side.

No treatment of other clinical patterns is allowed.

Main clinical inclusion criteria for subjects who did not participate in MRZ60201_3070_1:

* Female or male subject of 2 to 17 years age (inclusive).
* Uni- or bilateral CP with clinical need for BoNT injection to treat limb spasticity.
* AS score ≥ 2 in plantar flexors (at least unilaterally).
* Clinical need according to the clinical judgment of the investigator in one out of four treatment combinations:

  1. For LL(s) treatment only (Gross Motor Function Classification System [GMFCS] levels IV): Unilateral treatment of LL spasticity with 8 U/kg BW NT 201 (maximum of 200 U) into pes equinus, and 8 U/kg BW NT 201 (maximum of 200 U) into flexed knee or adducted thigh or bilateral treatment of LL spasticity with 8 U/kg BW NT 201 (maximum of 200 U) into each pes equinus (AS score ≥ 2 on both sides).
  2. For combined unilateral UL and unilateral LL, (GMFCS levels I-III): Unilateral treatment of LL spasticity with 8 U/kg BW NT 201 (maximum of 200 U) into pes equinus, and 8 U/kg BW NT 201 (maximum of 200 U) into flexed knee or adducted thigh plus Unilateral treatment of UL spasticity with 4 U/kg BW NT 201 (maximum of 100 U) into flexed elbow, flexed wrist, clenched fist, thumb in palm and/or pronated forearm.
  3. For combined unilateral UL and unilateral LL (GMFCS level IV-V): Unilateral treatment of LL spasticity with 8 U/kg BW NT 201 (maximum 200 U) into pes equinus, and 4 U/kg BW NT201 (maximum 100 U) into flexed knee or adducted thigh plus unilateral treatment of UL spasticity with 4 U/kg BW NT 201 (maximum of 100 U) into flexed elbow, flexed wrist, clenched fist, thumb in palm and/or pronated forearm.
  4. For combined unilateral UL and bilateral LL (GMFCS levels I-III): Bilateral treatment of LL spasticity with 8 U/kg BW NT 201 (maximum of 200 U) into each pes equinus (AS score ≥ 2 on both sides) plus unilateral treatment of UL spasticity with 4 U/kg BW NT 201 (maximum of 100 U) into flexed elbow, flexed wrist, clenched fist, thumb in palm and/or pronated forearm.

Exclusion Criteria:

Exclusion Criteria for subjects who completed MRZ60201_3070_1:

* Infection and/or inflammation in the area of the planned injection points.
* Pregnancy for female with history of menarche.
* Clinically relevant pathological findings indicating active disease of vital organs.

Exclusion Criteria for subjects who did not participate in MRZ60201_3070_1:

* Fixed contracture defined as severe restriction of the range of joint movement on passive stretch in the target clinical pattern(s) or predominant forms of muscle hypertonia other than spasticity (e.g., dystonia) in the target limb(s).
* Surgery in the pes equinus on side(s) intended to treat with BoNT injections within 12 months prior to Screening Visit (V1), within the screening period or planned for the time of participation in this study.
* Hip flexion requiring BoNT injection.
* Limitation of hip abduction to less than 40° or pre-diagnosed migrational percentage greater than 30.
* Vaccination within 2 weeks prior to Screening Visit (V1) and/or within the screening period.
* Non-resolved fractures of the treated limb.
* Ventilator dependency.
* Severe neurological diagnosis and comorbidity outside the spectrum of cerebral palsy.
* Pure dyskinetic CP or mixed CP with predominantly dyskinetic movements.
* Treatment with BoNT (other than study drug in this study) for any body region within 14 weeks prior to Screening Visit (V1), within the screening period and/or intended to be administered during the study period.
* Treatment with phenol or alcohol of any muscle within 6 months prior to Screening Visit (V1), within the screening period, and/or intended to be administered during the study period.
* Treatment with

  * drugs acting as peripheral muscle relaxants
  * intrathecal baclofen, or
  * oral anticoagulants administered within 2 weeks prior to Screening Visit (V1), within the screening period, and/or intended to be administered during the study period.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 370 (Actual)
Dates: Start 2013-08; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Merz Medical Expert, Study Director — Merz Pharmaceuticals GmbH
Locations (43):
- Merz Investigational Site #043036, Vienna, Austria
- Czechia (2):
  - Merz Investigational Site #420029, Brno
  - Merz Investigational Site #420028, Olomouc
- Estonia (2):
  - Merz Investigational Site #372001, Tallinn
  - Merz Investigational Site #372002, Tartu
- Germany (4):
  - Merz Investigational Site #049328, Bochum
  - Merz Investigational Site #049327, Munich
  - Merz Investigational Site #049329, Münster
  - Merz Investigational Site #049326, Vogtareuth
- Israel (3):
  - Merz Investigational Site #972003, Jerusalem
  - Merz Investigational Site #972001, Tel Aviv
  - Merz Investigational Site #972002, Tel Aviv
- Poland (7):
  - Merz Investigational Site #048089, Bialystok
  - Merz Investigational Site #048063, Gdansk
  - Merz Investigational Site #048059, Krakow
  - Merz Investigational Site #048084, Lublin
  - Merz Investigational Site #048072, Luboń
  - Merz Investigational Site #048075, Sandomierz
  - Merz Investigational Site #048061, Warsaw
- Romania (3):
  - Merz Investigational Site #040003, Bucharest
  - Merz Investigational Site #040001, Bucharest
  - Merz Investigational Site #040002, Iași
- Russia (6):
  - Merz Investigational Site #007014, Kazan'
  - Merz Investigational Site #007015, Khabarovsk
  - Merz Investigational Site #007018, Novosibirsk
  - Merz Investigational Site #007017, Saint Petersburg
  - Merz Investigational Site #007013, Smolensk
  - Merz Investigational Site #007019, Stavropol
- Slovakia (4):
  - Merz Investigational Site #421003, Banská Bystrica
  - Merz Investigational Site #421008, Bratislava
  - Merz Investigational Site #421006, Krompachy
  - Merz Investigational Site #421004, Levoča
- South Korea (4):
  - Merz Investigational Site #082019, Goyang
  - Merz Investigational Site #082021, Incheon
  - Merz Investigational Site #082018, Seongnam-si
  - Merz Investigational Site #082020, Seoul
- Turkey (Türkiye) (3):
  - Merz Investigational Site #090005, Elâzığ
  - Merz Investigational Site #090003, Izmir
  - Merz Investigational Site #090002, İzmit
- Ukraine (4):
  - Merz Investigational Site #380001, Dnipropetrovsk
  - Merz Investigational Site #380005, Kharkiv
  - Merz Investigational Site #380002, Kiev
  - Merz Investigational Site #380003, Odesa

REFERENCES:
- [Derived] Berweck S, Banach M, Gaebler-Spira D, Chambers HG, Schroeder AS, Geister TL, Althaus M, Hanschmann A, Vacchelli M, Bonfert MV, Heinen F, Dabrowski E. Safety Profile and Lack of Immunogenicity of IncobotulinumtoxinA in Pediatric Spasticity and Sialorrhea: A Pooled Analysis. Toxins (Basel). 2022 Aug 25;14(9):585. doi: 10.3390/toxins14090585. PMID 36136523

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 391 participants were screened, of which 370 participants were enrolled and treated. Of these, 124 participants were recruited from the lead-in study (62, 29 and 33 participants from the IncobotulinumtoxinA high, mid and low dose group respectively of study MRZ60201_3070_1 [2012-005054-30]) and 246 participants were newly recruited.
Groups:
- 16 - 20 U/kg Body Weight IncobotulinumtoxinA (Xeomin): Participants received total doses of 16 to 20 unit per kilogram (U/kg) body weight of IncobotulinumtoxinA (Xeomin) with a maximum of 400 to 500 units per injection treatment via intramuscular injection into spastic muscles on Day 1 of 4 treatment cycles (12 to 16 weeks treatment per each cycle). The higher dose could only be administered to participants with gross motor function classification system expanded and revised (GMFCS-E&R) levels I to III.
Period: Overall Study
Arm/Group | 16 - 20 U/kg Body Weight IncobotulinumtoxinA (Xeomin)
Started | 370
Completed | 319
Not Completed | 51
Not completed — Protocol Violation | 1
Not completed — Re-injection criteria not met; others | 13
Not completed — Physician Decision | 1
Not completed — Lack of Efficacy | 8
Not completed — Withdrawal by Subject | 20
Not completed — Adverse Event | 4
Not completed — Lost to Follow-up | 4

BASELINE CHARACTERISTICS:
Population: The safety evaluation set (SES) was the subset of all participants treated with investigational product (IP) at least once.
Groups:
- 16 - 20 U/kg Body Weight IncobotulinumtoxinA (Xeomin): Participants received total doses of 16 to 20 unit per kilogram (U/kg) body weight of IncobotulinumtoxinA (Xeomin) with a maximum of 400 to 500 units per injection treatment via intramuscular injection into spastic muscles on Day 1 of 4 treatment cycles (12 to 16 weeks treatment per each cycle). The higher dose could only be administered to participants with GMFCS-E&R levels I to III.
Arm/Group | 16 - 20 U/kg Body Weight IncobotulinumtoxinA (Xeomin)
Number analyzed (Participants) | 370
Age, Continuous [Mean (Standard Deviation); unit: years] | 6.2 (4.1)
Age, Customized [Count of Participants; unit: Participants]
  Children (2-11 years) | 317
  Adolescents (12-17 years) | 53
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 150
  Male | 220
Region of Enrollment [Number; unit: participants]
  Austria | 1
  South Korea | 59
  Romania | 22
  Turkey | 5
  Czechia | 1
  Ukraine | 170
  Poland | 67
  Israel | 1
  Slovakia | 5
  Germany | 1
  Estonia | 5
  Russia | 33

OUTCOME MEASURES:

1. Primary Outcome: Occurrence of Treatment Emergent Adverse Events (TEAEs) Overall and Per Injection Cycle
Description: TEAEs are events observed from the time point of first injection until end of study visit (Week 50-66). Values reported here refer to the number of participants affected.
Time Frame: From the timepoint of first injection up to end of study visit (Week 50-66)
Population: The SES was the subset of all participants treated with IP at least once.
Measure: Number; unit: participants
Arm/Group | 16 - 20 U/kg Body Weight IncobotulinumtoxinA (Xeomin)
Number analyzed (Participants) | 370
participants
  1st Injection Cycle | 53
  2nd Injection Cycle: number analyzed (Participants) | 350
  2nd Injection Cycle | 44
  3rd Injection Cycle: number analyzed (Participants) | 340
  3rd Injection Cycle | 26
  4th Injection Cycle: number analyzed (Participants) | 323
  4th Injection Cycle | 31
  Overall Period | 109

2. Primary Outcome: Occurrence of Treatment Emergent Adverse Events of Special Interest (TEAESI) Overall and Per Injection Cycle
Description: TEAEs occurring after treatment that were thought to possibly indicate toxin spread throughout the trial conduct are defined as TEAESI. Values reported here refer to the number of participants affected.
Time Frame: From the timepoint of first injection until end of study visit (Week 50-66)
Population: The SES was the subset of all participants treated with IP at least once.
Measure: Number; unit: participants
Arm/Group | 16 - 20 U/kg Body Weight IncobotulinumtoxinA (Xeomin)
Number analyzed (Participants) | 370
participants
  1st Injection Cycle | 1
  2nd Injection Cycle: number analyzed (Participants) | 350
  2nd Injection Cycle | 2
  3rd Injection Cycle: number analyzed (Participants) | 340
  3rd Injection Cycle | 1
  4th Injection Cycle: number analyzed (Participants) | 323
  4th Injection Cycle | 0
  Overall Period | 3

3. Primary Outcome: Occurrence of Treatment-emergent Serious Adverse Events (TESAEs) Overall and Per Injection Cycle
Description: TESAEs are events observed from the time point of first injection until end of study visit (Week 50-66). Values reported here refer to the number of participants affected.
Time Frame: From the timepoint of first injection until end of study visit (Week 50-66)
Population: The SES was the subset of all participants treated with IP at least once.
Measure: Number; unit: participants
Arm/Group | 16 - 20 U/kg Body Weight IncobotulinumtoxinA (Xeomin)
Number analyzed (Participants) | 370
participants
  1st Injection Cycle | 6
  2nd Injection Cycle: number analyzed (Participants) | 350
  2nd Injection Cycle | 5
  3rd Injection Cycle: number analyzed (Participants) | 340
  3rd Injection Cycle | 5
  4th Injection Cycle: number analyzed (Participants) | 323
  4th Injection Cycle | 1
  Overall Period | 16

4. Secondary Outcome: Investigator's Global Assessment of Tolerability at Day 99 (Week 14) of Each Injection Cycle
Description: The investigator's global assessment of tolerability was assessed on a 4-point ordinal scale where 1 = very good, 2 = good, 3 = moderate, and 4 = poor. Results for Day 99 (Week 14) of 4th injection cycles were collected at the end of study visit.
Time Frame: Day 99 (Week 14) of 1st, 2nd, 3rd and 4th injection cycle
Population: The SES was the subset of all participants treated with IP at least once.
Measure: Number; unit: participants
Arm/Group | 16 - 20 U/kg Body Weight IncobotulinumtoxinA (Xeomin)
Number analyzed (Participants) | 370
participants
  1st Injection Cycle: Very Good: number analyzed (Participants) | 350
  1st Injection Cycle: Very Good | 203
  1st Injection Cycle: Good: number analyzed (Participants) | 350
  1st Injection Cycle: Good | 119
  1st Injection Cycle: Moderate: number analyzed (Participants) | 350
  1st Injection Cycle: Moderate | 23
  1st Injection Cycle: Poor: number analyzed (Participants) | 350
  1st Injection Cycle: Poor | 5
  2nd Injection Cycle: Very Good: number analyzed (Participants) | 340
  2nd Injection Cycle: Very Good | 225
  2nd Injection Cycle: Good: number analyzed (Participants) | 340
  2nd Injection Cycle: Good | 87
  2nd Injection Cycle: Moderate: number analyzed (Participants) | 340
  2nd Injection Cycle: Moderate | 24
  2nd Injection Cycle: Poor: number analyzed (Participants) | 340
  2nd Injection Cycle: Poor | 4
  3rd Injection Cycle: Very Good: number analyzed (Participants) | 323
  3rd Injection Cycle: Very Good | 223
  3rd Injection Cycle: Good: number analyzed (Participants) | 323
  3rd Injection Cycle: Good | 74
  3rd Injection Cycle: Moderate: number analyzed (Participants) | 323
  3rd Injection Cycle: Moderate | 17
  3rd Injection Cycle: Poor: number analyzed (Participants) | 323
  3rd Injection Cycle: Poor | 9
  4th Injection Cycle: Very Good | 241
  4th Injection Cycle: Good | 76
  4th Injection Cycle: Moderate | 16
  4th Injection Cycle: Poor | 8
  4th Injection Cycle: Not assessed | 29

5. Secondary Outcome: Changes in AS Score of Left and Right Plantar Flexors (PF) From Baseline to All Other Visits, From Day 1 of Each Injection Cycle to Day 29 (Week 4), Day 57 (Week 8, 1st Injection Cycle Only) and Day 99 (Week 14) of the Respective Injection Cycle
Description: The Ashworth Scale (AS) is a well-known and commonly used scale in clinical trials with spasticity. In spastic muscles the resistance to passive movement is assessed. It is a 5-point scale that ranges from 0 (= no increase in tone) to 4 (=limb rigid in flexion or extension). For participants with bilateral pes equinus, the body side for efficacy analysis that is, "primary body side" was decided by investigator at screening and was kept throughout the entire study. V3 = Week 4 of 1st Injection Cycle; V4 = Week 8 of 1st Injection Cycle; V5 = Day 1 of 2nd Injection Cycle; V6= Week 4 of 2nd Injection Cycle; V7 = Day 1 of 3rd Injection Cycle; V8 = Week 4 of 3rd Injection Cycle; V9 = Day 1 of 4th Injection Cycle; V10 = Week 4 of 4th Injection Cycle; V11= Week 14th of 4th Injection Cycle = end of study visit.
Time Frame: Baseline (Day 1, Visit [V] 2) to all other visits (V3, V4, V5, V6, V7, V8, V9, V10, and V11); From Day 1 of Each Injection Cycle to Day 29 (Week 4), Day 57 (Week 8, 1st Injection Cycle only) and Day 99 (Week 14) of the respective Injection Cycle
Population: The full analysis set (FAS) was the subset of participants in the SES for whom at least a baseline value (Day 1 of the first cycle, Visit 2) of AS score of PF was available. For participants from lead-in study at least one post-baseline value was available.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 16 - 20 U/kg Body Weight IncobotulinumtoxinA (Xeomin)
Number analyzed (Participants) | 370
units on a scale
  Left PF Baseline (V2) to V3: number analyzed (Participants) | 302
  Left PF Baseline (V2) to V3 | -0.8 (0.7)
  Left PF Baseline (V2) to V4: number analyzed (Participants) | 304
  Left PF Baseline (V2) to V4 | -0.7 (0.7)
  Left PF Baseline (V2) to V5: number analyzed (Participants) | 288
  Left PF Baseline (V2) to V5 | -0.2 (0.5)
  Left PF Baseline (V2) to V6: number analyzed (Participants) | 288
  Left PF Baseline (V2) to V6 | -1.1 (0.8)
  Left PF Baseline (V2) to V7: number analyzed (Participants) | 282
  Left PF Baseline (V2) to V7 | -0.3 (0.6)
  Left PF Baseline (V2) to V8: number analyzed (Participants) | 281
  Left PF Baseline (V2) to V8 | -1.2 (0.8)
  Left PF Baseline (V2) to V9: number analyzed (Participants) | 268
  Left PF Baseline (V2) to V9 | -0.3 (0.6)
  Left PF Baseline (V2) to V10: number analyzed (Participants) | 268
  Left PF Baseline (V2) to V10 | -1.3 (0.8)
  Left PF Baseline (V2) to V11: number analyzed (Participants) | 282
  Left PF Baseline (V2) to V11 | -0.9 (0.8)
  Left PF 2nd Injection Cycle: Day 1 to Day 29: number analyzed (Participants) | 288
  Left PF 2nd Injection Cycle: Day 1 to Day 29 | -0.9 (0.8)
  Left PF 2nd Injection Cycle: Day 1 to Day 99: number analyzed (Participants) | 282
  Left PF 2nd Injection Cycle: Day 1 to Day 99 | -0.1 (0.4)
  Left PF 3rd Injection Cycle: Day 1 to Day 29: number analyzed (Participants) | 281
  Left PF 3rd Injection Cycle: Day 1 to Day 29 | -0.9 (0.7)
  Left PF 3rd Injection Cycle: Day 1 to Day 99: number analyzed (Participants) | 268
  Left PF 3rd Injection Cycle: Day 1 to Day 99 | -0.1 (0.4)
  Left PF 4th Injection Cycle: Day 1 to Day 29: number analyzed (Participants) | 268
  Left PF 4th Injection Cycle: Day 1 to Day 29 | -1 (0.7)
  Left PF 4th Injection Cycle: Day 1 to Day 99: number analyzed (Participants) | 264
  Left PF 4th Injection Cycle: Day 1 to Day 99 | -0.6 (0.7)
  Right PF Baseline (V2) to V3: number analyzed (Participants) | 306
  Right PF Baseline (V2) to V3 | -0.8 (0.7)
  Right PF Baseline (V2) to V4: number analyzed (Participants) | 308
  Right PF Baseline (V2) to V4 | -0.7 (0.7)
  Right PF Baseline (V2) to V5: number analyzed (Participants) | 293
  Right PF Baseline (V2) to V5 | -0.2 (0.5)
  Right PF Baseline (V2) to V6: number analyzed (Participants) | 291
  Right PF Baseline (V2) to V6 | -1 (0.8)
  Right PF Baseline (V2) to V7: number analyzed (Participants) | 285
  Right PF Baseline (V2) to V7 | -0.2 (0.5)
  Right PF Baseline (V2) to V8: number analyzed (Participants) | 284
  Right PF Baseline (V2) to V8 | -1.2 (0.8)
  Right PF Baseline (V2) to V9: number analyzed (Participants) | 273
  Right PF Baseline (V2) to V9 | -0.3 (0.5)
  Right PF Baseline (V2) to V10: number analyzed (Participants) | 273
  Right PF Baseline (V2) to V10 | -1.2 (0.8)
  Right PF Baseline (V2) to V11: number analyzed (Participants) | 287
  Right PF Baseline (V2) to V11 | -0.9 (0.8)
  Right PF 2nd Injection Cycle: Day 1 to Day 29: number analyzed (Participants) | 291
  Right PF 2nd Injection Cycle: Day 1 to Day 29 | -0.8 (0.7)
  Right PF 2nd Injection Cycle: Day 1 to Day 99: number analyzed (Participants) | 285
  Right PF 2nd Injection Cycle: Day 1 to Day 99 | -0.1 (0.4)
  Right PF 3rd Injection Cycle: Day 1 to Day 29: number analyzed (Participants) | 284
  Right PF 3rd Injection Cycle: Day 1 to Day 29 | -1 (0.7)
  Right PF 3rd Injection Cycle: Day 1 to Day 99: number analyzed (Participants) | 273
  Right PF 3rd Injection Cycle: Day 1 to Day 99 | 0 (0.4)
  Right PF 4th Injection Cycle: Day 1 to Day 29: number analyzed (Participants) | 273
  Right PF 4th Injection Cycle: Day 1 to Day 29 | -1 (0.7)
  Right PF 4th Injection Cycle: Day 1 to Day 99: number analyzed (Participants) | 270
  Right PF 4th Injection Cycle: Day 1 to Day 99 | -0.6 (0.7)

6. Secondary Outcome: Investigator's, Child's/Adolescent's, and Parent's/Caregiver's Global Impression of Change Scale (GICS) at Day 29 (Week 4) of Each Injection Cycle
Description: The GICS are global outcomes to assess the impression of change due to treatment. GICS were assessed by the investigator, by the participant (if feasible) and by parents'/caregiver (if applicable). GICS is 7-Point Likert Scale ranging from +3 (very much improved function) to -3 (very much worse function).
Time Frame: Day 29 (Week 4) of 1st, 2nd, 3rd and 4th injection cycle
Population: The FAS was the subset of participants in the SES for whom at least a baseline value (Day 1 of the first cycle, Visit 2) of AS score of PF was available. For participants from lead-in study at least one post-baseline value was available.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 16 - 20 U/kg Body Weight IncobotulinumtoxinA (Xeomin)
Number analyzed (Participants) | 370
units on a scale
  Investigator, Day 29 of 1st Injection Cycle: number analyzed (Participants) | 366
  Investigator, Day 29 of 1st Injection Cycle | 1.7 (0.7)
  Investigator, Day 29 of 2nd Injection Cycle: number analyzed (Participants) | 348
  Investigator, Day 29 of 2nd Injection Cycle | 1.8 (0.8)
  Investigator, Day 29 of 3rd Injection Cycle: number analyzed (Participants) | 339
  Investigator, Day 29 of 3rd Injection Cycle | 1.9 (0.8)
  Investigator, Day 29 of 4th Injection Cycle: number analyzed (Participants) | 323
  Investigator, Day 29 of 4th Injection Cycle | 2 (0.9)
  Participant, Day 29 of 1st Injection Cycle: number analyzed (Participants) | 124
  Participant, Day 29 of 1st Injection Cycle | 1.6 (0.8)
  Participant, Day 29 of 2nd Injection Cycle: number analyzed (Participants) | 117
  Participant, Day 29 of 2nd Injection Cycle | 1.7 (1)
  Participant, Day 29 of 3rd Injection Cycle: number analyzed (Participants) | 109
  Participant, Day 29 of 3rd Injection Cycle | 1.7 (0.9)
  Participant, Day 29 of 4th Injection Cycle: number analyzed (Participants) | 98
  Participant, Day 29 of 4th Injection Cycle | 1.8 (0.9)
  Parent/Caregiver, Day 29 of 1st Injection Cycle: number analyzed (Participants) | 366
  Parent/Caregiver, Day 29 of 1st Injection Cycle | 1.6 (0.8)
  Parent/Caregiver, Day 29 of 2nd Injection Cycle: number analyzed (Participants) | 348
  Parent/Caregiver, Day 29 of 2nd Injection Cycle | 1.8 (0.8)
  Parent/Caregiver, Day 29 of 3rd Injection Cycle: number analyzed (Participants) | 339
  Parent/Caregiver, Day 29 of 3rd Injection Cycle | 1.8 (0.8)
  Parent/Caregiver, Day 29 of 4th Injection Cycle: number analyzed (Participants) | 323
  Parent/Caregiver, Day 29 of 4th Injection Cycle | 1.9 (0.9)

7. Secondary Outcome: Investigator's Global Impression of Change of Plantar Flexor Spasticity Scale (GICS-PF) of Left and Right PF at Day 29 (Week 4) of Each Injection Cycle
Description: The GICS are global outcomes to assess the impression of change due to treatment. GICS were assessed by the investigator, by the participant (if feasible) and by parents'/caregiver (if applicable). GICS is a 7-Point Likert Scale ranging from +3 (very much improved function) to -3 (very much worse function). For participants with bilateral pes equinus, the body side for efficacy analysis that is "primary body side" was decided by investigator at screening and was kept throughout the entire study.
Time Frame: Day 29 (Week 4) of 1st, 2nd, 3rd and 4th injection cycle
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 16 - 20 U/kg Body Weight IncobotulinumtoxinA (Xeomin)
Number analyzed (Participants) | 370
units on a scale
  Left PF Day 29 of 1st Injection Cycle: number analyzed (Participants) | 302
  Left PF Day 29 of 1st Injection Cycle | 1.7 (0.7)
  Left PF Day 29 of 2nd Injection Cycle: number analyzed (Participants) | 288
  Left PF Day 29 of 2nd Injection Cycle | 1.8 (0.8)
  Left PF Day 29 of 3rd Injection Cycle: number analyzed (Participants) | 281
  Left PF Day 29 of 3rd Injection Cycle | 1.9 (0.8)
  Left PF Day 29 of 4th Injection Cycle: number analyzed (Participants) | 268
  Left PF Day 29 of 4th Injection Cycle | 2 (0.9)
  Right PF Day 29 of 1st Injection Cycle: number analyzed (Participants) | 306
  Right PF Day 29 of 1st Injection Cycle | 1.7 (0.7)
  Right PF Day 29 of 2nd Injection Cycle: number analyzed (Participants) | 291
  Right PF Day 29 of 2nd Injection Cycle | 1.8 (0.8)
  Right PF Day 29 of 3rd Injection Cycle: number analyzed (Participants) | 284
  Right PF Day 29 of 3rd Injection Cycle | 1.9 (0.8)
  Right PF Day 29 of 4th Injection Cycle: number analyzed (Participants) | 273
  Right PF Day 29 of 4th Injection Cycle | 2 (0.9)

8. Secondary Outcome: Changes in Modified Tardieu Scale (MTS) of Left and Right PF From Baseline to All Other Visits, From Day 1 of Each Injection Cycle (IC) to Day 29 (Week 4), Day 57 (Week 8, 1st IC Only) and Day 99 (Week 14) of the Respective Injection Cycle
Description: The MTS assesses spastic muscle tone by subtraction of two angles measured at different conditions of passive muscle stretch. R2 is the angle of passive range of motion with a passive movement at slow speed. R1 is the angle where a "catch-and-release" or clonus can be triggered at the fastest possible speed. Score values represent the measured (R2-R1) difference, that is, the dynamic tone component of the examined muscle(s). Decreases of (R2-R1) represent reductions in the dynamic component of spasticity, that is, improvement of dynamic muscle spasticity. V3 = Week 4 of 1st IC; V4 = Week 8 of 1st IC; V5 = Day 1 of 2nd IC; V6 = Week 4 of 2nd IC; V7 = Day 1 of 3rd IC; V8 = Week 4 of 3rd IC; V9 = Day 1 of 4th IC; V10 = Week 4 of 4th IC; V11 = Week 14 of 4th IC = end of study visit.
Time Frame: Baseline (Day 1, Visit [V] 2) to all other visits (V3, V4, V5, V6, V7, V8, V9, V10, and V11); From Day 1 of Each IC to Day 29 (Week 4), Day 57 (Week 8, 1st IC cycle only) and Day 99 (Week 14) of the respective IC
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | 16 - 20 U/kg Body Weight IncobotulinumtoxinA (Xeomin)
Number analyzed (Participants) | 370
Degrees
  Left PF Baseline(V2) to V3: number analyzed (Participants) | 302
  Left PF Baseline(V2) to V3 | -1.4 (10.6)
  Left PF Baseline (V2) to V4: number analyzed (Participants) | 304
  Left PF Baseline (V2) to V4 | -1.8 (9.8)
  Left PF Baseline (V2) to V5: number analyzed (Participants) | 288
  Left PF Baseline (V2) to V5 | -1 (7.1)
  Left PF Baseline (V2) to V6: number analyzed (Participants) | 288
  Left PF Baseline (V2) to V6 | -1 (12.3)
  Left PF Baseline (V2) to V7: number analyzed (Participants) | 282
  Left PF Baseline (V2) to V7 | -1.7 (8.1)
  Left PF Baseline (V2) to V8: number analyzed (Participants) | 281
  Left PF Baseline (V2) to V8 | -0.5 (13.8)
  Left PF Baseline (V2) to V9: number analyzed (Participants) | 268
  Left PF Baseline (V2) to V9 | -2.5 (8.1)
  Left PF Baseline (V2) to V10: number analyzed (Participants) | 268
  Left PF Baseline (V2) to V10 | -1.1 (14.6)
  Left PF Baseline (V2) to V11: number analyzed (Participants) | 283
  Left PF Baseline (V2) to V11 | -2.8 (10.9)
  Left PF 2nd IC: Day 1 to Day 29: number analyzed (Participants) | 288
  Left PF 2nd IC: Day 1 to Day 29 | 0 (11.1)
  Left PF 2nd IC: Day 1 to Day 99: number analyzed (Participants) | 282
  Left PF 2nd IC: Day 1 to Day 99 | -0.7 (5.8)
  Left PF 3rd IC: Day 1 to Day 29: number analyzed (Participants) | 281
  Left PF 3rd IC: Day 1 to Day 29 | 1.2 (10.9)
  Left PF 3rd IC: Day 1 to Day 99: number analyzed (Participants) | 268
  Left PF 3rd IC: Day 1 to Day 99 | -1 (5.8)
  Left PF 4th IC: Day 1 to Day 29: number analyzed (Participants) | 268
  Left PF 4th IC: Day 1 to Day 29 | 1.5 (11.7)
  Left PF 4th IC: Day 1 to Day 99: number analyzed (Participants) | 264
  Left PF 4th IC: Day 1 to Day 99 | 0 (7.9)
  Right PF Baseline (V2) to V3: number analyzed (Participants) | 306
  Right PF Baseline (V2) to V3 | -1.3 (10.6)
  Right PF Baseline (V2) to V4: number analyzed (Participants) | 308
  Right PF Baseline (V2) to V4 | -2.1 (9.3)
  Right PF Baseline (V2) to V5: number analyzed (Participants) | 293
  Right PF Baseline (V2) to V5 | -1.3 (7)
  Right PF Baseline (V2) to V6: number analyzed (Participants) | 291
  Right PF Baseline (V2) to V6 | -0.7 (12.4)
  Right PF Baseline (V2) to V7: number analyzed (Participants) | 285
  Right PF Baseline (V2) to V7 | -2.2 (8.3)
  Right PF Baseline (V2) to V8: number analyzed (Participants) | 284
  Right PF Baseline (V2) to V8 | -0.1 (13.9)
  Right PF Baseline (V2) to V9: number analyzed (Participants) | 273
  Right PF Baseline (V2) to V9 | -2.6 (8.5)
  Right PF Baseline (V2) to V10: number analyzed (Participants) | 273
  Right PF Baseline (V2) to V10 | -0.7 (14.4)
  Right PF Baseline (V2) to V11: number analyzed (Participants) | 287
  Right PF Baseline (V2) to V11 | -2.6 (11.7)
  Right PF 2nd IC: Day 1 to Day: number analyzed (Participants) | 291
  Right PF 2nd IC: Day 1 to Day | 0.6 (11.1)
  Right PF 2nd IC: Day 1 to Day 99: number analyzed (Participants) | 285
  Right PF 2nd IC: Day 1 to Day 99 | -1 (7.2)
  Right PF 3rd IC: Day 1 to Day 29: number analyzed (Participants) | 284
  Right PF 3rd IC: Day 1 to Day 29 | 2.1 (11.5)
  Right PF 3rd IC: Day 1 to Day 99: number analyzed (Participants) | 273
  Right PF 3rd IC: Day 1 to Day 99 | -0.5 (6.2)
  Right PF 4th IC: Day 1 to Day 29: number analyzed (Participants) | 273
  Right PF 4th IC: Day 1 to Day 29 | 1.9 (11.7)
  Right PF 4th IC: Day 1 to Day 99: number analyzed (Participants) | 270
  Right PF 4th IC: Day 1 to Day 99 | 0.4 (9.3)

9. Secondary Outcome: Change in Scores of Pain Intensity (From Participants) and Frequency (From Parent/Caregiver) From Baseline to All Visits, From Day 1 of Each IC to Day 29 (Week 4), Day 57 (Week 8, 1st IC Cycle Only) and Day 99 (Week 14) of Respective Injection
Description: The questionnaire on pain caused by Spasticity (QPS) is a participant-reported outcome for children and adolescents (2-17 years) with cerebral palsy on spasticity-related pain. Pain intensity (from participants) and pain frequency (from parent/caregiver) to be assessed with QPS. The QPS total score for pain intensity ranges from 0 ('No Hurt') to 10 ('Hurt Worst'). The QPS total score for the observed pain frequency ranges from 0 (Never) to 4 (Always). V3 = Week 4 of 1st IC; V4 = Week 8 of 1st IC; V5= Day 1 of 2nd IC; V6 = Week 4 of 2nd IC; V7 = Day 1 of 3rd IC; V8 = Week 4 of 3rd IC; V9 = Day 1 of 4th IC; V10 = Week 4 of 4th IC; V11 = Week 14 of 4th IC = end of study visit.
Time Frame: as for outcome 8
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 16 - 20 U/kg Body Weight IncobotulinumtoxinA (Xeomin)
Number analyzed (Participants) | 370
units on a scale
  Participants Baseline (V2) to V3: number analyzed (Participants) | 124
  Participants Baseline (V2) to V3 | -0.6 (1.7)
  Participants Baseline (V2) to V4: number analyzed (Participants) | 126
  Participants Baseline (V2) to V4 | -0.5 (2)
  Participants Baseline (V2) to V5: number analyzed (Participants) | 117
  Participants Baseline (V2) to V5 | -0.5 (1.7)
  Participants Baseline (V2) to V6: number analyzed (Participants) | 115
  Participants Baseline (V2) to V6 | -0.9 (1.9)
  Participants Baseline (V2) to V7: number analyzed (Participants) | 109
  Participants Baseline (V2) to V7 | -0.7 (1.7)
  Participants Baseline (V2) to V8: number analyzed (Participants) | 106
  Participants Baseline (V2) to V8 | -1.1 (1.9)
  Participants Baseline (V2) to V9: number analyzed (Participants) | 100
  Participants Baseline (V2) to V9 | -0.8 (1.7)
  Participants Baseline (V2) to V10: number analyzed (Participants) | 98
  Participants Baseline (V2) to V10 | -1.2 (2)
  Participants Baseline (V2) to V11: number analyzed (Participants) | 112
  Participants Baseline (V2) to V11 | -1 (1.8)
  Participants 2nd IC: Day 1 to Day 29: number analyzed (Participants) | 119
  Participants 2nd IC: Day 1 to Day 29 | -0.4 (1.4)
  Participants 2nd IC: Day 1 to Day 99: number analyzed (Participants) | 113
  Participants 2nd IC: Day 1 to Day 99 | -0.2 (1.2)
  Participants 3rd IC: Day 1 to Day 29: number analyzed (Participants) | 109
  Participants 3rd IC: Day 1 to Day 29 | -0.4 (1.2)
  Participants 3rd IC: Day 1 to Day 99: number analyzed (Participants) | 103
  Participants 3rd IC: Day 1 to Day 99 | -0.1 (0.9)
  Participants 4th IC: Day 1 to Day 29: number analyzed (Participants) | 101
  Participants 4th IC: Day 1 to Day 29 | -0.4 (1.3)
  Participants 4th IC: Day 1 to Day 99: number analyzed (Participants) | 101
  Participants 4th IC: Day 1 to Day 99 | -0.3 (1)
  Parent/Caregiver Baseline (V2) to V3: number analyzed (Participants) | 329
  Parent/Caregiver Baseline (V2) to V3 | -0.5 (0.8)
  Parent/Caregiver Baseline (V2) to V4: number analyzed (Participants) | 337
  Parent/Caregiver Baseline (V2) to V4 | -0.4 (0.8)
  Parent/Caregiver Baseline (V2) to V5: number analyzed (Participants) | 325
  Parent/Caregiver Baseline (V2) to V5 | -0.3 (0.8)
  Parent/Caregiver Baseline (V2) to V6: number analyzed (Participants) | 320
  Parent/Caregiver Baseline (V2) to V6 | -0.7 (0.9)
  Parent/Caregiver Baseline (V2) to V7: number analyzed (Participants) | 309
  Parent/Caregiver Baseline (V2) to V7 | -0.4 (0.9)
  Parent/Caregiver Baseline (V2) to V8: number analyzed (Participants) | 310
  Parent/Caregiver Baseline (V2) to V8 | -0.7 (1)
  Parent/Caregiver Baseline (V2) to V9: number analyzed (Participants) | 290
  Parent/Caregiver Baseline (V2) to V9 | -0.5 (0.9)
  Parent/Caregiver Baseline (V2) to V10: number analyzed (Participants) | 294
  Parent/Caregiver Baseline (V2) to V10 | -0.8 (1)
  Parent/Caregiver Baseline (V2) to V11: number analyzed (Participants) | 315
  Parent/Caregiver Baseline (V2) to V11 | -0.6 (0.9)
  Parent/Caregiver 2nd IC:Day 1 to Day 29: number analyzed (Participants) | 325
  Parent/Caregiver 2nd IC:Day 1 to Day 29 | -0.4 (0.7)
  Parent/Caregiver 2nd IC:Day 1 to Day 99: number analyzed (Participants) | 313
  Parent/Caregiver 2nd IC:Day 1 to Day 99 | -0.1 (0.6)
  Parent/Caregiver 3rd IC: Day 1 to Day 29: number analyzed (Participants) | 307
  Parent/Caregiver 3rd IC: Day 1 to Day 29 | -0.3 (0.7)
  Parent/Caregiver 3rd IC: Day 1 to Day 99: number analyzed (Participants) | 290
  Parent/Caregiver 3rd IC: Day 1 to Day 99 | -0.1 (0.5)
  Parent/Caregiver 4th IC: Day 1 to Day 29: number analyzed (Participants) | 288
  Parent/Caregiver 4th IC: Day 1 to Day 29 | -0.3 (0.7)
  Parent/Caregiver 4th IC: Day 1 to Day 99: number analyzed (Participants) | 286
  Parent/Caregiver 4th IC: Day 1 to Day 99 | -0.1 (0.6)

10. Secondary Outcome: Changes in Gross Motor Function Measure (GMFM)-66 Score From Baseline to All Injection Visits and End of Study
Description: The GMFM-66 is a standardized observational 66-item instrument designed and validated to measure change in gross motor function over time in participants with cerebral palsy. Score values represent the total GMFM-66 score. Total GMFM scores range from 0 (worst) to 100 (best).
Time Frame: Baseline to Day 1 of 2nd (V5), 3rd (V7), 4th (V9) IC and End of study (Week 44-68) (V11)
Population: The FAS was the subset of participants in the SES for whom at least a baseline value (Day 1 of the first cycle, Visit 2) of AS score of PF was available. For participants from lead-in study at least one post-baseline value was available. Therefore all participants from lead-in study were included in FAS.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 16 - 20 U/kg Body Weight IncobotulinumtoxinA (Xeomin)
Number analyzed (Participants) | 370
units on a scale
  Baseline (V2) to V5: number analyzed (Participants) | 349
  Baseline (V2) to V5 | 1.5 (3.2)
  Baseline (V2) to V7: number analyzed (Participants) | 340
  Baseline (V2) to V7 | 2.6 (4)
  Baseline (V2) to V9: number analyzed (Participants) | 322
  Baseline (V2) to V9 | 3.8 (5.1)
  Baseline (V2) to V11: number analyzed (Participants) | 339
  Baseline (V2) to V11 | 4.8 (5.9)

ADVERSE EVENTS:
Time Frame: From the time point of first injection up to end of study visit (Week 50-66)
Description: Adverse Events were collected systematically at each visit by the investigator.
Arm/Group | 16 - 20 U/kg Body Weight IncobotulinumtoxinA (Xeomin)
All-Cause Mortality (participants affected / at risk) | 0/370
Serious Adverse Events (participants affected / at risk) | 16/370
Other Adverse Events (participants affected / at risk) | 20/370
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 16 - 20 U/kg Body Weight IncobotulinumtoxinA (Xeomin) (N=370)
Tenotomy (Surgical and medical procedures) | 2 (3)
Cast application (Surgical and medical procedures) | 1 (1)
Arrhythmia (Cardiac disorders) | 1 (1)
Epilepsy (Nervous system disorders) | 2 (2)
Clonic convulsion (Nervous system disorders) | 1 (1)
Febrile convulsion (Nervous system disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (4)
Gastritis (Gastrointestinal disorders) | 1 (1)
Gastroenteritis (Infections and infestations) | 3 (4)
Bronchitis (Infections and infestations) | 2 (3)
Adenoiditis (Infections and infestations) | 1 (1)
Adenovirus infection (Infections and infestations) | 1 (2)
Croup infectious (Infections and infestations) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1)
Enteritis infectious (Infections and infestations) | 1 (1)
Respiratory tract infection viral (Infections and infestations) | 1 (1)
Hemagglutinin Type 1 and Neuraminidase Type 1 (H1N1) influenza (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 16 - 20 U/kg Body Weight IncobotulinumtoxinA (Xeomin) (N=370)
Nasopharyngitis (Infections and infestations) | 20 (34)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication of study information usually requires agreement with the sponsor. In case of justified doubts by the sponsor, the INVESTIGATOR will consider these doubts in the publication as long as the scientific neutrality is not affected.